CLINICAL TRIAL: NCT00374400
Title: The Paired Donation Consortium Paired Donation Program
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: The Paired Donation Consortium (Other)
Other Study IDs: PDC
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Transplant
Keywords: Kidney; Transplant; Paired donation; Living donor

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the protocol is to increase the number of living donor transplants by eliminating immune incompatibilities between donors and recipients through paired donation.

DETAILED DESCRIPTION:
The purpose of the protocol is to increase the number of living donor transplants by eliminating immune incompatibilities between donors and recipients through paired donation.

To increase the number of patients transplanted by paired donation by establishment of regional paired donation programs.

To develop educational programs for potential living donors and their recipient, as well as the opportunity for transplant professionals to increase acceptance of the PDC to maximize the opportunity for organ donation.

To identify and evaluate ethical and psychological factors that may influence the effects of paired donation on living kidney donation.

ELIGIBILITY:
Inclusion Criteria:

* Persons capable of providing written informed consent.
* Each recipient must have one or more medically suitable donors who are either ABO-incompatible or HLA-incompatible.

Exclusion Criteria:

* Persons with eligible, compatible donor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-09; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio